CLINICAL TRIAL: NCT02665689
Title: Influence of Diabetes Control on Treatment of Diabetic Macular Edema With Ranibizumab
Acronym: DORO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment pace was far below target.
Sponsor: Prof. Dr. Antonia M. Joussen (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Antonia M. Joussen, Prof. MD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DORO001
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Visual Acuity Reduced Transiently; Macular Edema, Cystoid
Keywords: Diabetic Macular Edema, Ranibizumab, Visual Acuity, Diabetic Control
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Observer-masking (assessment of BCVA, macular thickness, capillary drop-out) is done to guard against detection bias.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Glycemic Control (Active Comparator): Diabetic macular edema will be treated with 3 monthly ranibizumab (0,5mg) injections followed by PRN regimen. Patients randomized into this group will be controlled by their general practitioner or private diabetologist (usual care). The glycemic control (blood measurements of HbA1c) will be performed at trial site (Department of diabetology, endocrinology and nutritional medicine) every 3 months. The site will not influence or change the diabetes medication given by general physician and serves as an observer only to monitor the diabetic control.
  Interventions: Drug: ranibizumab
- Intensified Glycemic Control (Experimental): Diabetic macular edema will be treated with 3 monthly ranibizumab (0,5mg) injections followed by PRN regimen.
  Patients randomized into this group will be controlled at the trial site (Department of diabetology, endocrinology and nutritional medicine) during first year monthly, in the second study year every 3 months. The individual HbA1c will be targeted according to the general status reflecting other risk factors for the vasculopathy (e.g. BMI, smoking, blood pressure, lipid status). All effort will be done to reach the target blood pressure ≤ 140/90 mmHg and blood triglyceride level < 140 mg/dl: Further the patients will be educated to improve their eating habits in regard to reduce the carbohydrate intake.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Ranibizumab injections will be given for diabetic macular edema. In the experimental arm insulin injections and antihypertensiva will be applied.

SUMMARY:
The aim of the prospective randomized study is to investigate whether a intensified diabetic control program leads to better final visual acuity and less frequent diabetic ocular complications in patients with diabetic retinopathy when compared with a normal diabetic treatment.

DETAILED DESCRIPTION:
Patients with diabetic macular edema (DME) will be treated with intravitreal ranibizumab injections and the effect of optimal control of internal factors (eg. glycemia, blood pressure etc) on final functional (best corrected visual acuity-CBVA) and morphological (central retinal thickness-CRT) will be investigated. Patients will be randomized into two groups: Group with intensified diabetic control will be follow and investigated monthly at department of diabetology, endocrinology and nutritional medicine (Campus Benjamin Franklin) in Berlin with aim to reach the optimal glycemic control defined as HbA1c < 6,5%. Further, triglycerides values < 140 mg/dl and blood pressure < 140/90 mmHg will be pursued. Second group of patients will be followed by their general practitioner and in the study center only blood samples will be taken quarterly without active medical intervention.

BCVA, CRT and the number of required ranibizumab injections will we evaluated and compared between both study groups.

ELIGIBILITY:
Inclusion Criteria:

- Patients with diabetic macular edema relevant to visual acuity

* OCT central retinal thickness ≥ 250µm
* HbA1c > 6,5% at initial visit
* BCVA ≤0.8 and ≥0.05
* Age ≥18 years
* Written patient informed consent given

Exclusion Criteria:

* Previous treatment with intravitreal drugs in last 6 months
* Vitreous hemorrhage as a consequence of proliferative retinopathy
* Pregnancy
* Blood pressure of ≥ 180/100 (or uncontrolled pressures under pharmacological therapy)
* Chronic systemic or ocular inflammatory/autoimmune diseases (e.g. inflammatory bowel disease, Addison´s disease, Cushing Syndrome, Uveitis)
* Systemic cortisone or anti-VEGF therapy
* Acute systemic or ocular infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Charite, Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment has been stopped prematurely in August 2018 by the sponsor after the enrolment of four patients because the enrollment pace was far below target.
Pre-assignment Details: Screening period of seven days prior to randomization.
Period: Overall Study
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Trial termination | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of participants with history of ophthalmic disease [Count of Participants; unit: Participants] — Ophthalmic history features were collected (previous ophthalmic surgery, ocular trauma, glasses, glaucoma, glaucoma treatment, amblyopia, history of diabetic retinopathy).
  Participants | 2 | 2 | 4
Number of patients with medical history [Count of Participants; unit: Participants] — Medical history was determined (allergy, allergy medication, hypertonia, hypertonia medical compensation, hyperlipidemia, smoking, insulin treatment).
  Participants | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Difference of Best Corrected Visual Acuity Measured in ETDRS Letters Score Between Month 12 Baseline Visit
Description: Measured by the difference in ETDRS letters score between month 12 and baseline according to internal guideline of Charité department of ophthalmology.
Time Frame: Baseline to 12 months
Population: Of the four enrolled patients, only the two patients had 12-month visit. Since the time point for the evaluation of the primary endpoint was reached only for patients of study arm B, a comparison of both study arms was not possible and thus analysis of the primary endpoint was waived.
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Treatments With Ranibizumab up to 6, 12, 18 and 24 Months of Treatment
Description: For the number of treatments at 6, 12, 18 and 24 months, an ANOVA without any covariates was planned to be applied at each endpoint 6, 12, 18 and 24 months.
  As the time point 12 months for the evaluation of this secondary endpoint was reached only for patients of study arm B, a comparison of both study arms was not possible and thus statistical analysis of the endpoint was waived completely. None of the patients reached time points beyond month 12.
  Results are only shown descriptively. Ranibizumab injections were summed up per study arm as well as cumulative at each time point.
Time Frame: Baseline to 12 months
Population: At month 6, the two patients in study arm A had received six treatments each; the two patients in study arm B had received three and five treatments, respectively. At month 12, the two patients in study arm B had received three and six treatments, respectively. For none of the patients in study arm A, 12-month data was available.
Measure: Number; unit: Ranibizumab injections
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 2 | 2
Ranibizumab injections
  Month 6 | 12 | 8
  Month 12: number analyzed (Participants) | 0 | 2
  Month 12 |  | 9

3. Secondary Outcome: Difference of Best Corrected Visual Acuity Measured in ETDRS Letters Score Between Month 6, 12, 24 and Baseline Visit
Description: As the time point 12 months for the evaluation of this secondary endpoint was reached only for patients of study arm B, a comparison of both study arms was not possible and thus analysis of the endpoint was waived completely. Time point 24 months was reached by none of the patients due to trial discontinuation. Results are only shown descriptively.
  Best-corrected visual acuity (BCVA) score is shown as change in ETDRS letters score at the distinct time point compared to baseline. Higher scores mean a better outcome.
Time Frame: Baseline to 12 months
Population: BCVA score compared to baseline.
Measure: Number; unit: Letters improved
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 2 | 2
Letters improved
  Participant 1, month 6: number analyzed (Participants) | 1 | 0
  Participant 1, month 6 | 7 |
  Participant 2, month 6: number analyzed (Participants) | 1 | 0
  Participant 2, month 6 | 5 |
  Participant 3, month 6: number analyzed (Participants) | 0 | 1
  Participant 3, month 6 |  | 3
  Participant 4, month 6: number analyzed (Participants) | 0 | 1
  Participant 4, month 6 |  | 8
  Participant 3, month 12: number analyzed (Participants) | 0 | 1
  Participant 3, month 12 |  | 3
  Participant 4, month 12: number analyzed (Participants) | 0 | 1
  Participant 4, month 12 |  | 10

4. Secondary Outcome: Macular Thickness Change at 6, 12, 18 and 24 Months Compared to Baseline
Description: As the time point 12 months for the evaluation of this secondary endpoint was reached only for patients of study arm B, a comparison of both study arms was not possible and thus analysis of the endpoint was waived completely. None of the patients reached time points beyond month 12 due to trial discontinuation. Results are only shown descriptively.
  Macular thickness (study eye) is shown as change in thickness [µm] compared to individual baseline value. A reduction in thickness means improvement.
Time Frame: Baseline to 12 months
Population: For none of the patients in study arm A 12-month data was available. Time points beyond 6 months (18, 24 months) were reached by none of the patients due to trial discontinuation. Results are only shown descriptively.
Measure: Number; unit: µm
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 2 | 2
µm
  Participant 1, month 6: number analyzed (Participants) | 1 | 0
  Participant 1, month 6 | -91 |
  Participant 2, month 6: number analyzed (Participants) | 1 | 0
  Participant 2, month 6 | -319 |
  Participant 3, month 6: number analyzed (Participants) | 0 | 1
  Participant 3, month 6 |  | 10
  Participant 4, month 6: number analyzed (Participants) | 0 | 1
  Participant 4, month 6 |  | -103
  Participant 1, month 12: number analyzed (Participants) | 0 | 0
  Participant 2, month 12: number analyzed (Participants) | 0 | 0
  Participant 3, month 12: number analyzed (Participants) | 0 | 1
  Participant 3, month 12 |  | 23
  Participant 4, month 12: number analyzed (Participants) | 0 | 1
  Participant 4, month 12 |  | -101

5. Secondary Outcome: Time to Reach Target HbA1c
Time Frame: 24 months
Population: Originally, target HbA1c should have been defined individually for each patient by the investigator acc. to the patient's general status by risk factors for vasculopathy (Body-Mass-Index, smoking, blood pressure, lipid Status). However, definition of target HbA1c values was waived and only HbA1c values were documented (not shown here).
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Panretinal Laser Photocoagulation (PRP) Treatments Necessary for Neovascular Complications
Description: Need for PRP is up to the investigator's decision. Assessment was done on every visit.
  Intended time frame was baseline to 24 months. None of the patients reached time points beyond month 12 due to study discontinuation.
  Unit of measure is any separate investigator's decision to perform panretinal laser photocoagulation (PRP) for neovascular complications. Each PRP is counted separately.
Time Frame: Baseline to 12 months
Measure: Number; unit: number of PRPs across participants
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 2 | 2
number of PRPs across participants | 1 | 1

7. Secondary Outcome: Number of Participants With Retinal Detachment, Central Retinal Artery Occlusion, or Endophthalmitis and/or Ocular Adverse Events That Are Related to Treatment
Description: All ocular adverse events presented from baseline to 24 months will be documented.
Time Frame: Baseline to 12 months
Population: Patients in study arm A discontinued before month 12. None of the patients reached time points beyond month 12 due to trial discontinuation.
Measure: Number; unit: participants
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 2 | 2
participants
  Month 6 | 0 | 0
  Month 12: number analyzed (Participants) | 0 | 2
  Month 12 |  | 0

8. Secondary Outcome: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Description: All adverse events were documented. Causal relationship to study treatment was assessed by the investigators.
  Intended time frame was baseline to 24 months. None of the patients reached time points beyond 12 months due to study discontinuation.
Time Frame: Baseline to 12 months
Measure: Number; unit: participants
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
Number analyzed (Participants) | 2 | 2
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: First administration of the IMP until 30 days after the patient has stopped the treatment. Treatment is given individually acc. to summary of product characteristics following a pro re nata (as needed) scheme. Therefore adverse event data will be collected until time points individually for each patient but not longer than total trial duration (24 months). Time frame per protocol was baseline to 24 months. None of the patients reached time points beyond 12 months due to study discontinuation.
Arm/Group | Regular Glycemic Control | Intensified Glycemic Control
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regular Glycemic Control (N=2) | Intensified Glycemic Control (N=2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regular Glycemic Control (N=2) | Intensified Glycemic Control (N=2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 2 (2)
Heart valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injury associated with device (General disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Oedema peripheral (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Retinal exudates (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Anterior chamber disorder (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was stopped prematurely by the sponsor after enrolment of four patients since enrollment pace was far below target. Due to the limited number of patients, no conclusions in respect to the study aims can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02665689/Prot_SAP_000.pdf